CLINICAL TRIAL: NCT05618015
Title: Comparison of the Effectiveness of Supervised and Home-Based Progressive Resistant Training in the Mid-Term Postoperative Period in Female Total Knee Arthroplasty Patients
Brief Title: Comparison of the Supervised and Home-Based Progressive Resistant Training in Female Total Knee Arthroplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMMUHAN BAS ASLAN, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60116787-020/49018/13
Record Dates: First submitted 2022-11-07; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, it is not possible to blind participants or the treating physiotherapist. To reduce the bias risk, the outcome assessor was blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised progressive resistance training (Experimental): Supervised PRT was conducted face-to-face at the clinic
  Interventions: Procedure: Supervised progressive resistance training
- Home-based progressive resistance training (Active Comparator): Home-based PRT was conducted at home without supervision
  Interventions: Procedure: Home-based progressive resistance training

INTERVENTIONS:
Procedure: Supervised progressive resistance training — Exercises were performed with cable resistance training machine
  Arms: Supervised progressive resistance training
Procedure: Home-based progressive resistance training — In the first session, with the help of a physiotherapist, strengthening exercises were shown and taught to the patients. Two weeks after the beginning of the home-based PRT program, patients were called to check whether they were doing the exercises in the home program correctly. After the checking for exercise training, the patients were called by phone every two weeks for follow-up.
  Arms: Home-based progressive resistance training

SUMMARY:
Early postoperative rehabilitation programs after TKA aims to provide optimal functional recovery. The current rehabilitation process in TKA typically includes 2 to 3 months post-surgery, as the greatest declines in strength and functional performance occur immediately after surgery. Yet, the content, duration, and intensity of the rehabilitation programs for the reorganization of physical function after surgery have not yet been fully clarified. Whether home-based rehabilitation is comparable to supervised rehabilitation in the midterm period requires further research, as practices after TKA vary. The purpose of this study is to compare the effectiveness of supervised and home-based progressive resistance training (PRT) in the midterm postoperative period in female patients undergoing TKA.

DETAILED DESCRIPTION:
The objective of this study is to compare the pain, quadriceps strength, knee function, joint awareness, and quality of life between supervised or home-based PRT at 3 months after the total knee arthroplasty.

The study design is a single-blinded randomized trial. Both groups received standard physiotherapy for three months. In the third month postoperatively, supervised and home-based PRE, which consisted of sixteen sessions of exercise lasting eight weeks initiated. The clinical outcomes were compared at baseline (third month postoperatively) and the fifth month postoperative.

The clinical outcomes consisted of pain, range of motion (ROM), quadriceps and hip abductor muscle strength, and WOMAC (Western Ontario and McMaster University Arthritis Index ) score. The performance-based activity limitation test consisted of the 30-second sit-to-stand test, the 40-meter fast-paced walk test and the 9-step stair climb test. Joint awareness was assessed with Forgotten Joint Score-12 (FJS12). The quality of life was evaluated with the World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF).

ELIGIBILITY:
Inclusion Criteria:

* being a woman between the ages of 50-70
* underwent unilateral primary TKA surgery due to knee osteoarthritis three months ago
* understanding verbal and written instructions

Exclusion Criteria:

* revision TKA surgery
* neurological disease
* rheumatoid arthritis
* psychiatric problems
* severe limitation of knee ROM (knee flexion range < 90°)
* regular hypnotic or anxiolytics usage
* dementia.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Quadriceps and hip abductor muscles strength | 8 weeks
  The muscle strength was assessed with a hand-held dynamometer. For the quadriceps muscle test, the patient was seated on the edge of a hard bed. The dynamometer was placed on the midline of the tibia 5 cm proximal to the lateral malleolus. The patient was asked to force his leg into extension by overcoming the resistance of the dynamometer. For measurement of hip abductors muscle strength, the patient was placed supine and the dynamometer was placed on the lateral side of the leg, 5 cm proximal to the lateral malleolus. The patient was asked to force his leg into extension by overcoming the resistance of the dynamometer. The quadriceps and hip abductor muscles' strength were assessed at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
30s sit-to-stand test | 8 weeks
  The total number of sit-to-stand repetitions completed in 30 seconds was recorded. 30s sit-to-stand test is a measurement of lower limb strength and endurance. 30s sit-to-stand test was assessed at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
40m fast-paced walk test | 8 weeks
  The 40m fast-paced walking test measures short-distance walking activities. 40m fast-paced walk test was assessed at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
Stair climbing test | 8 weeks
  Functional limitations specific to ascending stairs were assessed with timed stair climbing and descending using a standard 9 steps (16-20 cm). Participants were instructed to climb stairs safely as soon as possible. Stair climbing test was assessed at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
Knee range of motion (ROM) | 8 weeks
  The universal goniometer was used to measure active knee flexion and extension while the participants were sitting with their knees hanging down on the edge of a firm bed. Knee ROM was assessed at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
Knee pain: Visual Analogy Scale (VAS) | 8 weeks
  Knee pain intensity during rest and activity (walking, sitting-to-standing, climbing stairs) were measured using separate 10 cm pain rating scale, with zero representing no pain at all and 10 representing worst imaginable pain. Knee pain was evaluated at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).

SECONDARY OUTCOMES:
The Western Ontario and McMaster University Osteoarthritis Index (WOMAC) | 8 weeks
  WOMAC was used to assess knee functions. WOMAC is a patient-reported, lower extremity-specific questionnaire and includes 24 questions: 17 on physical function, 5 on pain, and 2 on stiffness. WOMAC was evaluated at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
Fortgotten Joint Score-12 (FJS-12) | 8 weeks
  Artificial joint awareness was evaluated with FJS-12. The FJS-12 is a patient-reported outcome scale designed to assess joint awareness in the hips and knees. A five-point Likert response format consisting of a total of 12 questions, with a raw score converted from zero to 100 points, is used. FJS-12 was evaluated at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).
World Health Organization Quality of Life Instrument Short Form (WHOQOL-BREF) | 8 weeks
  Quality of life was evaluated with the World Health Organization Quality of Life Instrument, Short Form (WHOQOL-BREF). The WHOQOL-BREF questionnaire is a test used to evaluate the quality of life of healthy individuals and patients and consists of four subscales: physical health, psychological health, social relations and environmental areas. WHOQOL-BREF was evaluated at baseline (third month postoperatively) and after an 8-week intervention (fifth month postoperatively).

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan BAYRAK, PhD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jakobsen TL, Kehlet H, Husted H, Petersen J, Bandholm T. Early progressive strength training to enhance recovery after fast-track total knee arthroplasty: a randomized controlled trial. Arthritis Care Res (Hoboken). 2014 Dec;66(12):1856-66. doi: 10.1002/acr.22405. PMID 25074397
- [Result] Li D, Yang Z, Kang P, Xie X. Home-Based Compared with Hospital-Based Rehabilitation Program for Patients Undergoing Total Knee Arthroplasty for Osteoarthritis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2017 Jun;96(6):440-447. doi: 10.1097/PHM.0000000000000621. PMID 27584144
- [Result] Lopez-Liria R, Padilla-Gongora D, Catalan-Matamoros D, Rocamora-Perez P, Perez-de la Cruz S, Fernandez-Sanchez M. Home-Based versus Hospital-Based Rehabilitation Program after Total Knee Replacement. Biomed Res Int. 2015;2015:450421. doi: 10.1155/2015/450421. Epub 2015 Apr 16. PMID 25961017